CLINICAL TRIAL: NCT01066429
Title: Treatment With Infusional Dose-adjusted Etoposide/Vincristine/Doxorubicin/Bolus Cyclophosphamide/Dexamethasone and Rituximab (DA-EDOCH14-R) in Patients With Poor-prognosis Diffuse Large B-cell Lymphoma
Brief Title: DA-EDOCH14-R in Poor-prognosis Diffuse Large B-cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Principe de Asturias (Other)
Responsible Party: Hematology Service, Hospital Principe de Asturias
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DA-EDOCH14-R/07
Record Dates: First submitted 2010-02-08; First posted 2010-02-10 (Estimated); Last update posted 2010-02-12 (Estimated); Status verified 2009-12

CONDITIONS: Diffuse Large B-Cell Lymphoma (DLBCL)
Keywords: poor-prognosis diffuse large B-cell lymphoma; dose-adjusted; R-EDOCH-14; rituximab; age-adjusted IPI; toxicity
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Dexamethasone; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Poor prognosis DLBCL (No Intervention): Newly diagnosed patients with DLBCL and an age-adjusted IPI 2-3
  Interventions: Drug: Dexamethasone and dose-dense immunochemoterapy

INTERVENTIONS:
Drug: Dexamethasone and dose-dense immunochemoterapy — Administration every 14 days of the EDOCH-R scheme.
  Other Names: Dose-dense therapy; Rituximab; dexamethasone

SUMMARY:
Poor prognosis dufuse large B-cell lymphoma (DLBCL) represents 50% of all DLBCL with overall cure rates ranging from 50-60% with modern dose-dense immunochemotherapy regimens such as R-CHOP14. Using an alternative strategy, as infusional and dose-adjusted R-EPOCH, the investigators have shown an 83% of complete responses (CR), with an estimated 5-year overall survival (OS) rate of 75% (García-Suárez et al. British Journal of Haematology 2007, 136:276). Despite this improvement in outcome, the search for new treatment strategies should continue. Therefore, compared with prior R-EPOCH the investigators decided to investigate whether the introduction of dexamethasone (40 mg IV on days 1-5) in place of prednisone (based upon data which demonstrated that the former was associated with enhanced Central Nervious System penetration) and the reduction of treatment intervals from 3 to 2 weeks would be feasible and might improve the outcome in this group of patients.

DETAILED DESCRIPTION:
Medication, Dose and Method for Administration:

* Rituximab: 375 mg/m2, endovenous, according to the protocol of the service, day 1 (except in the first cycle, in which it will be on day 5).
* Etoposide: 50 mg/m2/day, in continuous 24-hour infusion, days 1 to 4.
* Adriamycin: 10 mg/m2/day, in continuous 24-hour infusion of, days 1 to 4.
* Vincristine: 0.4 mg/m2/day, in continuous 24-hour infusion, days 1 to 4
* Dexamethasone: 40 mg, endovenous, days 1 to 5. Followed by prednisone 30 mg (day +6), 20 mg (day +7), and 10 mg (day +8).
* Cyclophosphamide: 750 mg/m2, endovenous, in 30 minutes, day 5, after ending the continuous infusion of adriamycin, etoposide and vincristine.
* MESNA (If the dose of Cyclophosphamide is > 1 g/m2

ELIGIBILITY:
Inclusion Criteria:

* Signing the Informed Consent.
* Histology: diffuse large B-cell lymphoma de novo (primary mediastinal B-cell lymphomas will be included provided that they have a mass greater than 7 cm in larger diameter) and follicular NHL grade 3b.
* aaIPI: 2-3.
* Age: Between 18 and 70 years.
* General Condition (ECOG/WHO): Proper organic function, defined by: FEVI ≥ 40%, serum creatinine < 150 µmol/L, serum bilirubin < 30 µmol/L, control of other medical conditions such as: infection, leukocytes ≥ 3.5 x 109/l and platelets ≥ 100 x 109/l (except if they are caused by lymphomatous infiltration of bone marrow or of the spleen).

Exclusion Criteria:

* HIV-positive.
* Pregnancy or breastfeeding.
* Serious disease compromising the performance of the therapeutic regimen.
* Recent history of another malignant disease (except skin cancer different from melanoma or carcinoma in-situ of the cervix), prior radiotherapy or chemotherapy, history of indolent lymphoma.
* CNS infiltration at diagnosis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
efficacy of the EDOCH14-R scheme at an adjusted dose | Between December 2009 and January 2012

SECONDARY OUTCOMES:
hematological and extra-hematological toxicity of the EDOCH14-R scheme | Between december 2009 and January 2012

CONTACTS AND LOCATIONS:
Overall Officials: Julio Garcia-Suarez, MD, PhD, Principal Investigator — Service of Hematology, Principe de Asturias University Hospital,
Locations (1):
- Principe de Asturias University Hospital, Alcalá de Henares, Madrid, Spain

REFERENCES:
- [Derived] Garcia-Suarez J, Flores E, Callejas M, Arribas I, Gil-Fernandez JJ, Olmedilla G, Curto N, Guillen H, Casco CR, Martin Y, Burgaleta C. Two-weekly dose-adjusted (DA)-EPOCH-like chemotherapy with high-dose dexamethasone plus rituximab (DA-EDOCH14-R) in poor-prognostic untreated diffuse large B-cell lymphoma. Br J Haematol. 2013 Feb;160(4):510-4. doi: 10.1111/bjh.12144. Epub 2012 Dec 11. PMID 23228045